CLINICAL TRIAL: NCT05283993
Title: A Prospective Cohort Study of Patients With Plasma Cell Disorders (PCDs) in PKUFH
Brief Title: A Cohort Study of Plasma Cell Disorders (PCDs) in PKUFH
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yujun DONG, chief of department of hematology, Peking University First Hospital
Other Study IDs: PekingUFHH
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma; Amyloidosis; Cryoglobulinemia; Castleman's Disease; Light Chain Deposition Disease; Heavy Chain Deposition Disease; Polyneuropathy Organomegaly Endocrinopathy Monoclonal Gammopathy and Skin Changes; Smoldering Multiple Myeloma; Plasma Cell Leukemia; Monoclonal Gammopathy of Undetermined Significance (MGUS); Monoclonal Gammopathy of Renal Significance (MGRS); Monoclonal Gammopathy of Neurological Significance (MGNS)
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis; Cryoglobulinemia; Castleman Disease; POEMS Syndrome; Smoldering Multiple Myeloma; Leukemia, Plasma Cell; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood, bone marrow aspirate and urine samples will be banked for future research involving adults with PCDs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The primary aim is to establish a prospective cohort of patients with plasma cell disorders (PCDs). All of the hospitalized PCD patients who are willing to sign the informed consent form (ICF) will be included in this study. Clinical characteristics, treatment options and responses will be collected. Peripheral blood, bone marrow aspirate and urine samples before and after the treatment will banked for future research. Our team will focus on the clinical and pathological features of PCDs, the correlation between the minimal residual disease (MRD) status and prognosis, and the role of Tumor Microenvironment (TME) in the pathogenesis and progress of PCDs.

DETAILED DESCRIPTION:
Primary

1. To establish a prospective cohort of patients with PCDs in PKUFH.
2. To dynamically analyze the relation between MRD status and prognosis, and the possible role of TME in PCD patients.

Secondary To collect peripheral blood, bone marrow aspirate and urine samples from PCD patients for future study, such as the tumor clone selection and evolution.

OUTLINE: PCD patients enrolled in this study will be assessed at baseline, clinical and laboratory data and biological samples be collected. Follow-up will be done at the 1, 3, 6, 12 months and then yearly after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included are those with confirmed diagnosis of PCDs and hospitalized into Peking University First Hospital (PKUFH)
2. Patients of plasma cell disorders (PCDs) are recruited. PCDs include monoclonal gammopathy of uncertain significance; smoldering myeloma; multiple myeloma; plasma cell leukemia; amyloidosis; light chain deposition disease; heavy chain deposition disease; Castleman's disease (CD); Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal gammopathy and Skin changes syndrome; cryoglobulinemia; Monoclonal Gammopathy of Renal Significance (MGRS); Monoclonal gammopathy of neurological significance (MGNS).
3. Patients are included into this cohort after signing the ICFs.

Exclusion Criteria:

Significant comorbidity may be life-threatening.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with confirmed diagnosis of PCDs will be enrolled. PCDs include monoclonal gammopathy of uncertain significance; smoldering myeloma; multiple myeloma; plasma cell leukemia; amyloidosis; light chain deposition disease; heavy chain deposition disease; Castleman's disease (CD); Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal gammopathy and Skin changes syndrome; cryoglobulinemia; Monoclonal Gammopathy of Renal Significance (MGRS); Monoclonal gammopathy of neurological significance (MGNS).
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
A Cohort Study of Plasma Cell Disorders (PCDs) in PKUFH | 10 years
  To measure the treatment response in the cohort study of PCDs in PKUFH.The treatment response is done according to the criteria of the International Myeloma Working Group (IWMG) of 2016.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China